CLINICAL TRIAL: NCT06704529
Title: Cortical Processing of Proprioception Related to Pitching Performance in Baseball Players With Glenohumeral Internal Rotation Deficit
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202407026RINB
Record Dates: First submitted 2024-08-21; First posted 2024-11-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Glenohumeral Internal Rotation Deficit
Keywords: proprioception; baseball; pitching performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- baseball players with GIRD
  Interventions: Behavioral: pitching motion
- baseball players without GIRD
  Interventions: Behavioral: pitching motion

INTERVENTIONS:
Behavioral: pitching motion — participants pitch fastball to the strike zone

SUMMARY:
The current study aims to characterize the cortical activity and proprioceptive acuity in baseball players with glenohumeral internal rotation deficit (GIRD). Additionally, the correlations between cortical activity, proprioceptive acuity, and pitching performance will be examined. The evaluation of proprioception will be conducted using the active joint reposition sense of the shoulder. Simultaneously, the investigators will record cortical activity by electroencephalography (EEG). To represent pitching performance, the investigators will collect ball velocity and pitching accuracy. This will help the investigators understand the process of proprioception in the central nervous system, as well as factors associated with pitching performance in baseball players with GIRD.

ELIGIBILITY:
Inclusion Criteria:

* playing baseball for at least one year
* still active in training or competition
* frequency of training or games should be at least 3 hours per week

Exclusion Criteria:

* current dominant upper extremities pain
* a history of upper extremities surgical interventions or fractures or dislocation or degenerative joint disease
* cervical radiculopathy within 6 months
* lower extremities injury or surgery within the current 6 months
* Visual analog scale (VAS) > 5 during movement in the experiment

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: GIRD is defined as 20° less GH IR ROM in the dominant shoulder compared to the non-dominant shoulder. Players without GIRD will be recruited to match the characteristics and sports involvement data (age ±3 years, right-handed or left-handed, pitcher or fielder, practice time >10 hours/week or <10 hours/week, baseball experience >3 years or <3 years) of the GIRD players.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Active joint reposition test | baseline
  Participants will mimic the pitching motion with reducing the influence from the lower limb by kneeling the knee and hip of the nondominant side 90° and their foot are flat on the ground. They will be blindfolded, with their non-throwing hand resting on the thigh. The reproducing arm-cocking and ball-release positions will be tested at random sequences for six trials, respectively. Results or feedback regarding the accuracy of individual trials will not be provided at any time. The acuity of active joint reposition will be calculated by 3-dimensional variable error scores for scapulothoracic (internal-external rotation, upward-downward rotation, posterior-anterior tilt) and glenohumeral (internal-external rotation, horizontal abduction-adduction, abduction-adduction) joint 55. Three-dimensional variable error scores (3DVE) reflect acuity (measured in degrees) in all planes of motion measured for individual joints.
Pitching performance | baseline
  Pitching performance will be collected by radar gun (JUGS company, Tualatin, OR, USA) and digital camera (JVC GC-PX100B, Yokohama, Japan) for ball velocity and pitching location, respectively. Participants will pitch on a mound 18.44 m away from the home plate. The target will be aligned with the theoretical line extending from the right edge of the home plate at a height of approximately 30 cm above the ground.
  After warming up at their own pace, each participant throws 30 game-like effort pitches in three 10-pitch sessions without specific instruction on focusing their attention. The fastest velocity of 10 pitches will be collected for analysis.

SECONDARY OUTCOMES:
Shoulder range of motion | baseline
  The tester grasps the subject's forearm in a supine position to measure the shoulder horizontal adduction/abduction. The humerus will be moved until the movement ceases (firm end-feel), indicating the end of shoulder tissue flexibility. The recorder places the digital inclinometer parallel to the humerus. Each measurement will be performed 3 times, and the average data will be analyzed.
  GH internal/external (IR/ER) ranges will be measured accordingly following the method in a previous study. Participants lay down supine with 90° shoulder abduction and elbow flexion. Then GH IR/ER will be measured by the main assessor using a digital inclinometer by stabilizing the scapula by grasping the coracoid process and the spine of the scapula posteriorly, then moving the forearm to reach the end range. Each measurement will be performed 3 times, and the average data will be used for analysis.
Humeral retrotorsion | baseline
  Humeral retrotorsion will be measured with the T3300 ultrasound system (BenQ, Taipei, Taiwan). Participants lay supine with 90° shoulder abduction and elbow flexion. The main assessor places the transducer on the participant's anterior shoulder for a short-axis view of the lesser and greater tubercles. The two-person technique is adopted. The first assessor adjusts the probe perpendicular to the floor and rotates the participant's humerus with a line connecting the greater and lesser tubercles parallel to the horizontal plane. Then, the second assessor places a digital inclinometer on the ulnar side of the forearm to record the rotation angle, which is defined as the humeral retroversion.23 The ICC3,k of intra-rater reliability is 0.995. Each measurement will be performed 3 times, and averaged data will be used for analysis.
Acromiohumeral distance | baseline
  Acromiohumeral distance will be measured with the ultrasound transducer placed on the lateral aspect of the acromion in line with the longitudinal axis of the humerus to visualize the shortest distance between the humerus and the acromion.58 Three consecutive ultrasound images of the acromiohumeral distance are captured. The investigator captures 3 more consecutive ultrasound images at rest while the participant sit with the shoulder in the neutral position. The shortest distance will be measured with built-in calipers. The ICC3,k for intra-rater reliability is 0.963. Each measurement will be performed 3 times and averaged data will be used for analysis.
Rotator cuff thickness | baseline
  The probe will be positioned on the bicipital grove horizontally to measure subscapularis tendon thickness in a short axis of view. The participant's forearm is placed with the elbow flexed to 90° in slight internal rotation, with the palm facing upward and medially. This position allows the bicipital groove to be brought to an anterior position, allowing clear visualization of the tendon within the grove. .
Posterior capsule thickness | baseline
  For measurement of the posterior capsule thickness, the participants sit upright in a chair with both forearms resting on the thighs and upper arms by the participant's sides. The examiner positions a transducer on the posterior shoulder and visualizes the glenoid labrum, humeral head, rotator cuff, and posterior capsule. The posterior capsule is defined as the tissue immediately lateral to the tip of the labrum between the humeral head and rotator cuff. When the capsule is identified in the image, posterior capsule thickness will be measured with built-in calipers. The ICC3,k for intra-rater reliability is 0.951. Each measurement will be performed 3 times, and averaged data will be used for analysis.
Kerlan-Jobe Orthopaedic Clinic Shoulder and Elbow score (KJOC) | baseline
  The KJOC is the most common questionnaire for overhead athletes, and it was conducted in several studies.66 Recently, the Major League Baseball (MLB) organization adopted this evaluation tool as the standard for recovering injuries in MLB players.67 The questionnaire is commonly used to assess shoulder function and performance. It is valid, reliable in its pilot form, and responsive to the tested population of adult overhead athletes.66 KJOC questionnaire ranges from 0 to 100, and the lower score represents a limited function.
Posterior capsule elasticity | baseline
  To measure the posterior capsule elasticity, the participants sit upright in a chair with both forearms resting on the thighs and upper arms by the participant's sides. The examiner positions a transducer on the posterior shoulder and visualizes the glenoid labrum, humeral head, rotator cuff, and posterior capsule. The posterior capsule is defined as the tissue immediately lateral to the tip of the labrum between the humeral head and rotator cuff. When the capsule is identified in the image, posterior capsule elasticity will be recorded. Each measurement will be performed 3 times and averaged data will be used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Background] Mine K, Nakayama T, Milanese S, Grimmer K. Effectiveness of Stretching on Posterior Shoulder Tightness and Glenohumeral Internal-Rotation Deficit: A Systematic Review of Randomized Controlled Trials. J Sport Rehabil. 2017 Jul;26(4):294-305. doi: 10.1123/jsr.2015-0172. Epub 2016 Aug 24. PMID 27632891
- [Background] Aldridge R, Stephen Guffey J, Whitehead MT, Head P. The effects of a daily stretching protocol on passive glenohumeral internal rotation in overhead throwing collegiate athletes. Int J Sports Phys Ther. 2012 Aug;7(4):365-71. PMID 22893856
- [Background] Johnson JE, Fullmer JA, Nielsen CM, Johnson JK, Moorman CT 3rd. Glenohumeral Internal Rotation Deficit and Injuries: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2018 May 22;6(5):2325967118773322. doi: 10.1177/2325967118773322. eCollection 2018 May. PMID 29845083
- [Background] Meister K, Day T, Horodyski M, Kaminski TW, Wasik MP, Tillman S. Rotational motion changes in the glenohumeral joint of the adolescent/Little League baseball player. Am J Sports Med. 2005 May;33(5):693-8. doi: 10.1177/0363546504269936. Epub 2005 Feb 16. PMID 15722284
- [Background] Freehill MT, Archer KR, Diffenderfer BW, Ebel BG, Cosgarea AJ, McFarland EG. Changes in collegiate starting pitchers' range of motion after single game and season. Phys Sportsmed. 2014 Feb;42(1):69-74. doi: 10.3810/psm.2014.02.2049. PMID 24565823
- [Background] Astolfi MM, Struminger AH, Royer TD, Kaminski TW, Swanik CB. Adaptations of the Shoulder to Overhead Throwing in Youth Athletes. J Athl Train. 2015 Jul;50(7):726-32. doi: 10.4085/1062-6040-50.1.14. Epub 2015 Mar 26. PMID 25811844